CLINICAL TRIAL: NCT06327243
Title: The Effects of Kinesio Taping on Knee Pain, Range of Motion, and Functional Performance in People With Knee Osteoarthritis
Brief Title: The Effects of Kinesio Taping on Pain, Range of Motion, and Functional Performance in People With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taibah University (Other)
Responsible Party: Principal Investigator, Marwan Mahmoud Aljohani, Assistant professor, Taibah University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TUMRHS
Record Dates: First submitted 2024-03-12; First posted 2024-03-25 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Athletic Tape

STUDY DESIGN:
Intervention Model Description: In a randomized and single-blinded approach, participants are divided into two groups. One group receives actual Kinesio taping, while the other undergoes a sham procedure, with neither group aware of their specific treatment type to ensure unbiased results.
Who Masked: Participant
Masking Description: Participants will not know if they are receiving the actual Kinesio Taping (KT) treatment or a sham taping. The KT will be applied following the correct standards for the rectus femoris muscle, including appropriate stretching. Conversely, the placebo taping will be applied horizontally across the muscle fibers without any stretching. The therapists applying the tape will know which treatment each participant is allocated to ensure that the application of either the real KT or the placebo taping aligns with the study's protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kineso taping group (Experimental)
  Interventions: Other: Elastic tape ( kinesio tape)
- Sham group (Sham Comparator)
  Interventions: Other: Sham Taping

INTERVENTIONS:
Other: Elastic tape ( kinesio tape) — This group will receive the tape on their quadriceps femoris muscle. First, the tape will be cut in a Y-shaped Kinesio type and then applied over the quadriceps femoris muscle. The tape will be applied at a point of 5 cm inferior to the anterior superior iliac spine to the patella (origin to insertion), with the patient in a supine position with 25% tension on the tape. Then, each patient will flex his or her knee, and the Y-shaped tape (the end of the tape) will be circled around the patella, ending at its inferior side with no tension.
  Arms: Kineso taping group
Other: Sham Taping — Sham taping will be applied horizontally across the muscle fibers without any stretching. the tape here will be applied transverse to the quadriceps femoris muscle. The patients will be in a supine position with their hips flexed at 30 degrees and their knees flexed at 60 degrees.
  Arms: Sham group

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of Kinesio Taping in individuals with knee osteoarthritis (KOA). KOA is a common condition that can lead to pain, stiffness, and decreased mobility. The main questions it aims to answer are:

* Does Kinesio Taping reduce pain in individuals with KOA?
* Can Kinesio Taping improve the range of motion and functional performance in those suffering from KOA?

Participants will be asked to:

Attend assessment sessions at the outpatient Physical Therapy clinic at Taibah University.

Undergo Kinesio Taping three times over 12 days. Complete specific physical tests and questionnaires before and after the intervention period to measure their pain and mobility.

Researchers will compare the group that receives Kinesio Taping with the group that receives sham (placebo) taping to see if there are significant differences in pain reduction and improvements in movement and daily function.

DETAILED DESCRIPTION:
Study Overview

This clinical trial explores Kinesio Taping's (KT) effect on knee osteoarthritis (KOA) in adults. It delves into whether KT can alleviate pain and improve joint movement and daily functioning. The research, hosted at Taibah University's Physical Therapy clinic, focuses on practical benefits for patients with KOA, a condition that leads to significant discomfort and mobility issues, especially prevalent in Saudi Arabia.

Study Design

In a randomized and single-blinded approach, participants are divided into two groups. One group receives actual Kinesio taping, while the other undergoes a sham procedure, with neither group aware of their specific treatment type to ensure unbiased results.

Intervention Procedures

Participants undergo three Kinesio taping sessions spread over 12 days. The taping technique is performed according to prescribed methods that target the quadriceps femoris muscle, believed to influence pain perception and joint function positively.

The study employs a before-and-after intervention assessment model. Initial data collection includes patients' demographic details and baseline characteristics related to their health status and disease severity. Following the intervention, the same measures are reassessed to evaluate any changes attributed to the KT.

ELIGIBILITY:
Inclusion Criteria:

* Patients clinically and radiologically diagnosed with unilateral or bilateral knee OA.
* Independent gait
* Any grade on the Kellgren-Lawrence scale

Exclusion Criteria:

* Previous fractures of the femur and/or tibia.
* Comorbidities such as neurological diseases, malnutrition, and other inflammatory and/or infectious diseases.
* Radicular pain in the lower limbs or diabetic neuritis.
* Prior physiotherapy in the past month.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-09 (Actual)

PRIMARY OUTCOMES:
Pain (Visual analog scale) | At baseline (pre-intervention), and then repeated immediately after the intervention
  a tool that measures pain intensity. It consists of a straight line, typically 10 cm long, with "no pain" on one end and "severe pain" on the other. Participants mark a point on the line that represents their current level of pain, providing a quantitative measure of pain intensity.
Knee range of motion | At baseline (pre-intervention), and then repeated immediately after the intervention
  the knee range of motion measured by goniometer
Timed up and go test | At baseline (pre-intervention), and then repeated immediately after the intervention
  measures mobility by timing how long it takes a person to stand up from a chair, walk 3 meters, turn around, walk back, and sit down. Longer times suggest decreased mobility and a higher fall risk.
The 50-foot Walk | At baseline (pre-intervention), and then repeated immediately after the intervention
  measures walking speed over a short distance. Participants walk 50 feet as quickly and safely as possible, and the time taken is recorded. This test assesses functional mobility and endurance.
Knee Osteoarthritis Outcome Score (KOOS) | At baseline (pre-intervention), and then repeated immediately after the intervention
  is a patient-reported questionnaire developed to assess the patient's opinion about their knee and associated problems. It consists of five subscales: Pain, Other Symptoms, Function in daily living (ADL), Function in Sport and Recreation (Sport/Rec), and knee-related Quality of Life (QOL). The scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems. It is widely used in the assessment of the short-term and long-term consequences of knee osteoarthritis.

CONTACTS AND LOCATIONS:
Overall Officials: Marwan MA Aljohani, Phd, Principal Investigator — Taibah University
Locations (1):
- Taibah University, Madinah, Saudi Arabia